CLINICAL TRIAL: NCT01420367
Title: Are Post-operative Antibiotics Indicated in Simple Appendicitis? a Prospective Randomized Trial
Brief Title: Are Post-operative Antibiotics Indicated in Simple Appendicitis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Monash Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U1111-1123-7877
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2011-08

CONDITIONS: Appendicitis
Keywords: Paediatric; Simple; Non-perforated
MeSH Terms: conditions — Appendicitis; Charcot-Marie-Tooth disease, Type 1C | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose of antibiotics (Experimental): This group will receive one dose of IV metronidazole (12.5mg/kg up to 500mg) and cefazolin (25mg/kg up to 1g) in the pre-operative period and two post-operative IV 'doses' of normal saline 8 and 16 hours after the pre-operative dose, which will act as a placebo and facilitate blinding.
  Interventions: Drug: metronidazole and cephalzolin
- Three doses of antibiotics (Active Comparator): This group will receive one pre-operative dose of IV metronidazole (12.5mg/kg up to 500mg) and cefazolin (25mg/kg up to 1g) and two post-operative doses of IV metronidazole (12.5mg/kg up to 500mg) and cefazolin (25mg/kg up to 1g) 8 and 16 hours after the pre-operative dose.
  Interventions: Drug: metronidazole and cephalzolin

INTERVENTIONS:
Drug: metronidazole and cephalzolin — IV doses of metronidazole (12.5mg/kg up to 500mg) and cefazolin (25mg/kg up to 1g). One dose for study arm, two for comparative arm.

SUMMARY:
Hypothesis: A single dose of prophylactic antibiotics is as effective as a three dose regime in preventing post-operative complications in paediatric patients with simple appendicitis.

This project will compare patients 16 years and under with simple appendicitis (appendicitis that is not perforated or gangrenous). Patients will be randomly divided into two groups;

* Group one will receive a single pre-operative dose of antibiotics (metronidazole 12.5mg/kg up to 500mg and cefazolin 25mg/kg up to 1g) and two 'doses' of normal saline (placebo) eight and sixteen hours after the initial dose, respectively.
* Group two will receive one pre-operative dose of antibiotics (metronidazole 12.5mg/kg up to 500mg and cefazolin 25mg/kg up to 1g) and two post-operative doses, eight and sixteen hours after the first dose, respectively.

Group allocation will be concealed from the patient and their guardian, the treating surgical team and outcome assessors (triple blinded). A process to rapidly reveal group allocation if required will be in place.

The aim of the study is to determine if a single dose of antibiotics is as effective as three doses in preventing post-operative infection. This will be assessed by comparing:

* Duration of hospital stay from operation until discharge, based on a standardised discharge criteria.
* Development of wound infection or requirement of antibiotics in the six weeks post-operation
* Need for re-admission.

Information will be collected prospectively from each patient's hospital notes and from a follow-up phone call six weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have their appendix removed and are found on operation to have 'simple appendicitis' as defined in the Cochrane review[7]. That is an appendix that is non-inflamed, acutely inflamed, phlegmonous, suppurative or mildly inflamed.

Exclusion Criteria:

* Patients who on operation are found to have 'complicated appendicitis' defined as an appendix that is gangrenous or perforated.
* Patients who pre-operatively appear to be acutely septic or for another reason require extended antibiotic therapy.
* Patients who, at operation, are found to have other pathology e.g. Meckel's Diverticulum, Intussusception; requiring surgical or medical intervention.
* Any patient whose guardian does not wish for them to participate in the study.
* Patients who have additional co-morbidities, including diabetes, immuno-suppression, cardiac, renal or liver failure.
* If the child continues to show sign of sepsis, in terms of fever, tachycardia, he/she will be discontinued from the study and be given additional doses of antibiotics, as clinically indicated.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Presence of post-operative infection in the six weeks following appendectomy | 6 weeks
  Defined by wound infection, fever (>38.5) or evidence of sepsis.
Requirement of further antibiotic therapy in the six weeks following appendectomy | 6 weeks
  Administration of antibiotics either by hospital or general practitioner in the 6 week post-operative period.

SECONDARY OUTCOMES:
Time to discharge taken from the time of operation to the time the child first satisfied the discharge criteria | 1 week
  Discharge criteria:
  Pain adequately controlled with oral analgesia Tolerating full diet Afebrile
Re-admission in the six weeks following appendectomy | 6 weeks
  Re-admission to the treating hospital or any other hospital in the 6 weeks post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Mennie, MBBS, Principal Investigator — Monash University; Wei Cheng, MBBS, Study Director — Monash Medical Centre
Locations (1):
- Monash Medical Centre, Clayton, Victoria, Australia